CLINICAL TRIAL: NCT06405178
Title: Sodium-Glucose Co-Transporter-2 Inhibitors as Adjuvant Therapy With Letrozole in Induction of Ovulation in Women With Polycystic Ovarian Syndrome
Brief Title: Adjuvant Therapy With Letrozole in Induction of Ovulation With Polycystic Ovarian Syndrome
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, principle investigator/Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Xigiduo PCO
Record Dates: First submitted 2024-05-04; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Polycystic Ovary
Keywords: Sodium-Glucose Co-Transporter-2 Inhibitors; Letrozole; Ovulation; Polycystic Ovarian Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; dapagliflozin; Letrozole

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Metformin 1000mg (Experimental)
  Interventions: Drug: Metformin; Drug: Letrozole
- Dapagliflozin 10mg (Experimental)
  Interventions: Drug: Dapagliflozin; Drug: Letrozole
- Dapagliflozin-Metformin 10/1000mg (Experimental)
  Interventions: Drug: Dapagliflozin/Metformin; Drug: Letrozole
- control group. (No Intervention)

INTERVENTIONS:
Drug: Metformin — Insulin Sensitizer
  Other Names: Glucophage 1000
  Arms: Metformin 1000mg
Drug: Dapagliflozin — Sodium-Glucose Co-transporter-2
  Other Names: Forxiga
  Arms: Dapagliflozin 10mg
Drug: Dapagliflozin/Metformin — Anti diabetic drug
  Other Names: Xigduo
  Arms: Dapagliflozin-Metformin 10/1000mg
Drug: Letrozole — Aromataze inhibitor
  Other Names: femara
  Arms: Dapagliflozin 10mg; Dapagliflozin-Metformin 10/1000mg; Metformin 1000mg

SUMMARY:
The aim of the study is to assess the efficacy of adjuvant therapy dapagliflozin, metformin as monotherapy and combination of both in comparison to control group in induction of ovulation with letrozole in women PCOS, focusing specifically on rates of ovulation and pregnancy.

DETAILED DESCRIPTION:
The study will be a randomized controlled clinical trial. Once the eligibility from screening visit is determined prior to baseline visit, randomization will be made by computer randomization for women who are admitted to Beni-Suef University Hospital.

* Before initiation of the study, the population will be divided randomly into 4 equal groups: group A, B, C and D. The adjuvant therapy of each group will be group (A) Metformin 1000mg, group (B) Dapagliflozin 10mg, Group(C) Combined Dapagliflozin-Metformin 10/1000mg and group (D) with no adjuvant therapy (control group).
* The adjuvant therapy will be taken once daily with a main meal and started one month before initiation of letrozole. All groups will take letrozole 2.5mg twice daily from the third day of the cycle for 5 days.

This treatment regimen will continue for three cycles unless positive pregnancy is achieved. No diet restriction will be recommended during the study or change in the lifestyle. The population will be asked to inform about any side effects that may happen during the study. A written informed consent will be obtained from each woman participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* PCOS will based on European Society of Human Reproduction and Embryology/American Society for Reproductive Medicine (ESHRE/ASRM) criteria, the diagnosis is made when at least two of the following criteria are met:

  * oilgo and/or anovulation (infrequent or no ovulation),
  * clinical and/or biochemical signs of hyperandrogenism including hirsutism, acne and/or increased testosterone levels
  * polycystic ovaries on ultrasound (defined as those containing at least 12 follicles measuring 2-9 mm in diameter arranged peripherally around an echo-dense stroma and/or with increased ovarian volume of at least 10 ml).

Exclusion Criteria:

* Other causes of hyperandrogenism mimic PCOS such as congenital adrenal hyperplasia, Cushing's syndrome, or androgen secreting tumors are excluded.
* Persistent hyperprolactinemia,
* thyroid dysfunction defined as TSH < 0.2 mIU/ML or >5.5 mIU/mL)
* patients with menopausal levels of FSH (> 15 mIU/mL) (A normal level within the last year is adequate for enter the study).
* Liver disease is defined as AST or ALT > 2 times normal or total bilirubin >2.5 mg/dL, #kidney disease defined as BUN > 30 mg/dL or serum creatinine> 1.4 mg/dL or significant

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Pregnancy | 3 cycles ( 3 months / one month for each cycle)
  Serum HCG positive

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Beni-Suef University, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No